CLINICAL TRIAL: NCT00189150
Title: Pharmacokinetics of Mycophenolate Mofetil Alone and in Combination With Valganciclovir in Renal and Heart Transplant Recipients
Brief Title: Pharmacokinetics of Mmf and Valganciclovir
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Hoffmann-La Roche (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Val060
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2016-05

CONDITIONS: Kidney Transplant Recipient; Heart Transplant Recipient
Keywords: Valganciclovir; Mycophenolate Mofetil; Pharmacokinetic; Interaction; MPA
MeSH Terms: interventions — Mycophenolic Acid; Valganciclovir

INTERVENTIONS:
Drug: Mycophenolate mofetil
Drug: Valganciclovir

SUMMARY:
The primary objective of this study is to determine whether a clinically significant PK drug interaction ( a 30% difference in the AUC of MPA) exists between mycophenolate mofetil (under steady state conditions) and VGCV in renal and cardiac transplant recipients.

This study will provide clinically relevant information to the transplant community. It will more clearly delineate whether a clinically significant PK drug interaction exists between mycophenolate mofetil (under steady-state conditions)and VGCV. Given the established dose/efficacy relationship of both MMF and VGCV, this study will provide improved dosing guidelines and potentially avoid adverse outcomes due to empiric dosage adjustments.

DETAILED DESCRIPTION:
Mycophenolate mofetil (immunosuppressant, MMF) and valganciclovir (antiviral, VGCV) are commonly administered together in transplant patients. Following oral administration, both MMF and VGCV are metabolized to active forms, mycophenolic acid (MPA) and gancoclovir (GCV) respectively. Both MPA and GCV are eliminated through kidney and renal excretion, but there is no data on how MPA pharmacokinetic parameters are affected by GCV at steady state condition. Both MPA and GCV can cause neutropenia and although unsubstantiated, some clinicians have observed an increased occurrence of neutropenia when these agents are used in combination. In the presence of neutropenia, practitioners are often challenged when making decisions regarding whether the dosage of one or both agents should be reduced. It would be useful to know whether the neutropenia is due to increased drug concentration or whether it is due to direct effects of these agents on the bone marrow.

ELIGIBILITY:
Inclusion Criteria:

The subject must be able to give informed consent for the study. Stable renal or cardiac transplant patients age 18 years and older. Patients must not have had an acute rejection episode within the previous 30 days of the 1st PK study.

Renal transplant patients with serum creatinine < 2 mg/dL and with change in serum creatinine < 25% within the 2 weeks prior to the 1st PK study.

Renal and cardiac transplant patients receiving VGCV for prophylaxis of CMV while concomitantly receiving MMF.

Stable MMF dose: the dose of MMF must not have been adjusted within 1 week of the 1st PK study and must be the same during the 2nd PK study Stable renal function during the study period (change in serum creatinine < 25%)

Exclusion Criteria:

Patients who are not prescribed MMF maintenance therapy or are receiving Myfortic.

Patients who do not require VGCV prophylaxis (CMV negative recipients of CMV negative donor organs).

Patients who have their MMF doses adjusted either < 1 week before the 1st scheduled PK study or anytime during the study period.

Patients whose serum creatinine changes by > 25% within 2 weeks prior to study initiation.

Patients whose hematocrit < 28%. Patients who received other organ transplants in addition to a kidney or heart. Patients who are pregnant or breast-feeding. Patients prescribed bile acids, bile acid sequestrants, potassium binding resins, or magnesium/aluminum-containing antacids.

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2005-04; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
To determine whether a clinically significant pharmacokinetic drug interaction exists between mycophenolate mofetil and valganciclovir under steady state conditions in renal and heart transplant recipients

SECONDARY OUTCOMES:
To determine whether the effects of valganciclovir on mycophenolate mofetil pharmacokinetic parameters are different between renal and heart transplant recipients

CONTACTS AND LOCATIONS:
Overall Officials: Jeong M Park, MS, PharmD, Principal Investigator — University of Michigan Hospital
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States